CLINICAL TRIAL: NCT00528814
Title: Effect of a School Based Hand Sanitizer Program on Asthma
Brief Title: Effectiveness of a School-Based Hand Sanitizer Program on Reducing Asthma Exacerbations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blue Cross Blue Shield (Other); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 519; R01HL086972 (NIH)
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Asthma
Keywords: Hand Sanitizer; Respiratory Infection
MeSH Terms: conditions — Asthma; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Two Step Hand-Hygiene (Experimental): Hand washing plus hand sanitizer
  Interventions: Other: Active Hand Sanitizer
- Usual Care Hand Hygiene (No Intervention)

INTERVENTIONS:
Other: Active Hand Sanitizer — Active Hand Sanitizer
  Other Names: Purell
  Arms: Two Step Hand-Hygiene

SUMMARY:
Asthma is a common, serious illness among children in the United States. Improving hand cleanliness and hygiene may prevent the spread of viruses that can cause asthma exacerbations. This study will evaluate the effectiveness of a school-based hand sanitizer program at reducing the frequency of exacerbations in children with asthma.

DETAILED DESCRIPTION:
In the United States, almost 9 million children have been diagnosed with asthma. It is a leading cause of hospitalizations and school absenteeism among children. Asthma symptoms are often seasonal, with the greatest number of exacerbations occurring in autumn and the fewest in mid-summer. Elementary school children are the most vulnerable to these seasonal changes, and many children experience an increase in exacerbations at the beginning of the school year. Recent research suggests that this seasonal peak in exacerbations is primarily caused by viral respiratory tract infections that are spread among children in school. Regular handwashing has been widely recognized as the most effective way to stop the spread of viruses and infectious illnesses. However, effective handwashing methods among school-age children can be inconsistent. Time constraints, a frequent lack of soap and towels, inconveniently located sinks, and water-saving faucets are all barriers to thorough handwashing. Improving hand hygiene through the use of antimicrobial rinse-free hand sanitizers in school classrooms may be a simple and effective way to reduce the risk of transmitting viruses that can cause asthma exacerbations. The purpose of this study is to evaluate the effectiveness of a school-based hand sanitizer program at decreasing exacerbations in children with asthma.

This study will enroll children with asthma who are attending one of the 32 participating schools. Each school will be randomly assigned to either use their usual hand hygiene practices in Year 1, followed by a two-step hand hygiene program including hand washing plus hand sanitizer in Year 2, or vice versa. Each participant will log in to an Internet-based data collection system on a daily basis to document their asthma symptoms and peak flow meter readings. Teachers will also log in daily to verify participants' data and to document participants' absences and the reason for the absence. Quick relief medication use will be recorded and measured through the use of a Doser device on participants' inhalers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with asthma
* Enrolled in a participating elementary school

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 527 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbations | Measured at Years 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: William Bailey, MD, Principal Investigator — University of Alabama at Birmingham, Lung Health Center
Locations (1):
- University of Alabama at Birmingham, Lung Health Center, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Gerald LB, Gerald JK, Zhang B, McClure LA, Bailey WC, Harrington KF. Can a school-based hand hygiene program reduce asthma exacerbations among elementary school children? J Allergy Clin Immunol. 2012 Dec;130(6):1317-24. doi: 10.1016/j.jaci.2012.08.031. Epub 2012 Oct 12. PMID 23069487
- [Derived] Gerald LB, Gerald JK, McClure LA, Harrington K, Erwin S, Bailey WC. Redesigning a large school-based clinical trial in response to changes in community practice. Clin Trials. 2011 Jun;8(3):311-9. doi: 10.1177/1740774511403513. PMID 21730079